CLINICAL TRIAL: NCT00035334
Title: A Phase II/III Study of the Safety and Efficacy of NC-503 in Patients Suffering From Secondary (AA) Amyloidosis
Brief Title: Study of the Safety and Efficacy of NC-503 in Secondary (AA) Amyloidosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bellus Health Inc. - a GSK company (Industry)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-503004; NCT00017667 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-02-14 (Estimated); Status verified 2006-02

CONDITIONS: Secondary (AA) Amyloidosis; Rheumatoid Arthritis; Nephrotic Syndrome; Familial Mediterranean Syndrome; Kidney Diseases; Gastrointestinal Diseases
Keywords: Familial Mediterranean Fever; Amyloidosis; Secondary (AA) Amyloidosis; Nephrotic Syndrome
MeSH Terms: conditions — Neoplasm Metastasis; Amyloidosis; Arthritis, Rheumatoid; Nephrotic Syndrome; Kidney Diseases; Gastrointestinal Diseases; Familial Mediterranean Fever | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: NC-503 (Anti-amyloidotic (AA) Agent)

SUMMARY:
The main objective of this study is to evaluate the safety and efficacy of NC-503 compared to placebo in patients with secondary (AA) amyloidosis using a composite assessment of clinical improvement/worsening of both renal and gastrointestinal functions.

DETAILED DESCRIPTION:
AA amyloidosis is associated with chronic inflammatory conditions (rheumatoid arthritis, ankylosing spondylitis, inflammatory bowel disease), chronic infection (tuberculosis, osteomyelitis), and Familial Mediterranean Fever. Rheumatoid arthritis is the major cause of AA amyloidosis in Western Europe and North America. The most common clinical feature of AA amyloidosis is renal dysfunction manifested as nephrotic-range proteinuria or renal insufficiency at the time of diagnosis. End-stage renal failure is the cause of death in 40-60% of cases. Gastrointestinal involvement is also frequent and is usually manifested as chronic diarrhea, body weight loss and malabsorption. Enlargement of the liver and spleen may also occur in some patients. The median survival time from diagnosis varies from 2 to 8 years depending on the stage of the disease at time of diagnosis. The goal of the current therapy in AA amyloidosis is the control of the associated disease. However, the current approaches for the treatment of AA amyloidosis are unspecific, toxic, invasive, and not sufficiently effective in many cases. NC-503 was specifically designed to compete with the naturally occurring sulfated GAGs for the binding to amyloidogenic precursor proteins, and to inhibit amyloid deposition into tissues. The proposed therapy with NC-503 is based on the prevention of the amyloid fibril formation. The objective of this clinical phase II/III study is to determine the efficacy and safety of NC-503 compared to a placebo in patients suffering from secondary (AA) amyloidosis by the assessment of clinical improvement/ worsening of both renal and gastrointestinal functions.

ELIGIBILITY:
PROTOCOL INCLUSION CRITERIA

* Patients must be 18 years of age or older.
* Males and females. If women of childbearing potential (i.e., not surgically sterilized or post-menopausal greater than one year) the patient must be using effective birth control.
* Diagnosis of AA amyloidosis demonstrated by positive biopsy (Congo red staining) and immunohistochemistry or immunoelectron microscopy at screening visit. Tissue from previous biopsy can be used for confirmation of diagnosis, if available.
* Persistent proteinuria defined as urinary protein excretion ? 1g/24h in two distinct 24-h urine collections at least 1 week apart within 3 months prior to study entry (baseline, Month 0 visit) without evidence of urinary tract infection or overt heart failure (NYHA class III or more); OR creatinine clearance ? 60 mL/min in two distinct measures at least 1 week apart within 3 months prior to study entry (baseline, Month 0 visit).
* Creatinine clearance ? 20 mL/min AND serum creatinine ? 3 mg/dl within 3 months prior to study entry (baseline, Month 0 visit).
* Written informed consent.

PROTOCOL EXCLUSION CRITERIA

* Evidence or suspicion of renal or renovascular diseases other than renal AA amyloidosis.
* Presence of diabetes mellitus (Type I and II).
* Evidence of a cause of potentially reversible reduced renal function, such as accelerated hypertension or drug nephrotoxicity.
* AST, ALT, or ALP > 5 times the upper limit of normal, or total bilirubin 50% above upper limits of normal.
* Presence of any other clinically significant diseases that could interfere with the interpretation of study results or compromise patient safety or any conditions that could reduce life expectancy to less than two years.
* Use of an investigational drug within thirty days prior to the screening visit.
* Active alcohol and/or drug abuse.
* Initiation of or any changes in ACE inhibitor therapy within 3 months prior to the screening visit.
* Initiation of or any changes in cytotoxic agents/colchicine therapy within 3 months prior to the screening visit.
* Inability to provide legal consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-10; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (26):
- United States (4):
  - Indiana University School of Medicine, Department of Pathology and Laboratory Medicine,, Indianapolis, Indiana
  - Boston Medical Center, Renal Division, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
- Rheumatism Foundation Hospital, Heinola, Finland
- France (3):
  - Centre Hospitalier du Mans, Service de Rhumatologie, Le Mans
  - Hôpital Claude Huriez, Service de médecine Interne, Clinique Médicale A, Lille
  - Hôpital Cochin, Centre de Recherche et d'Explorations Fonctionnelles, Paris
- Israel (2):
  - Bnai Zion Medical Center, Haifa
  - Heller Institute of Medical Research, Sheba Medical Center, Tel Litwinsky
- Italian Group for Systemic Amyloidosis, Biotechnology Research Laboratories, IRCCS Policlinico San Matteo, Internal Medicine and Medical Oncology, Pavia, Italy
- Vilnius University Hospital, Vilnius, Lithuania
- University Hospital Groningen, Department of Medicine, Division of Rheumatology, Groningen, Netherlands
- Poland (2):
  - Instytut Reumatologiczny, Warsaw
  - Okregowy Szpital Kolejowy, Zaklad Reumatologii, Wroclaw
- Russia (2):
  - Institute of Rheumatology RAMS, Moscow
  - Regional Hospital No. 1, Yekaterinburg
- Spain (4):
  - Hospital Universitario Germans Trias I Pujol, Servicio de Reumatologia, Badalona
  - Hospital Clinic I Provincial de Barcelona, Jefe del Departamento de Reumatologia, Barcelona
  - Ciutad Sanitària y Universitària de Bellvitge, Servicio de Reumatologia, Hospitalet de Llobregat, Llobregat
  - Hospital Clinico San Carlos de Madrid, Servicio de Reumatologia, Madrid
- Turkey (Türkiye) (3):
  - Cerrehpasa Tip Fakultesi, Askaray, Istanbul, Turkey
  - Istanbul Faculty of Medicine, Department of Internal Medicine, Division of Rheumatology, Istanbul
  - Marmara University Medical School Hospital, Department of Rheumatology, Uskudar, Altunizade, Istanbul
- United Kingdom (2):
  - Royal Free and University College Medical School, Department of Medicine, National Amyloidosis Centre, London
  - Gartnavel General Hospital, Scotland

REFERENCES:
- [Background] Safety, Tolerability and Pharmacokinetic Profile of FibrillexTM (Anti-AA Amyloid Agent) in Healthy and Renal Impaired Subjects. Garceau D., Gurbindo C., Laurin J. Neurochem Inc. Reference: Proceedings from the IXth International Symposium on Amyloidosis , 2001 (Budapest, Hungary)
- [Derived] Dember LM, Hawkins PN, Hazenberg BP, Gorevic PD, Merlini G, Butrimiene I, Livneh A, Lesnyak O, Puechal X, Lachmann HJ, Obici L, Balshaw R, Garceau D, Hauck W, Skinner M; Eprodisate for AA Amyloidosis Trial Group. Eprodisate for the treatment of renal disease in AA amyloidosis. N Engl J Med. 2007 Jun 7;356(23):2349-60. doi: 10.1056/NEJMoa065644. PMID 17554116